CLINICAL TRIAL: NCT05008731
Title: Effect of Botulinum Toxin on Hamstring Contracture and the Occurrence of Cyclops Syndrome After Anterior Cruciate Ligament Reconstruction
Brief Title: Cyclops Syndrome After Anterior Cruciate Ligament Reconstruction
Acronym: SCALA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-005742-42
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hamstring Contractures
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomised, double-blind study of two parallel groups of 66 patients with post-reconstruction ACL hamstring contracture treated with an ultrasound-guided injection at two points on the body of the hamstring
  * Group 1: botulinum toxin: 100 units (0.5ml) in 1 injection
  * Group 2: placebo: 0.5 ml in 1 injection
Who Masked: Participant, Investigator
Masking Description: A placebo is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): botulinum toxin: 100 units (0.5ml) in 1 injection
  Interventions: Drug: Botulinum toxin
- Group 2 (Placebo Comparator): Placebo: 0.5 ml in 1 injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Botulinum toxin — 100 units (0.5ml) in 1 injection
  Arms: Group 1
Other: Placebo — Placebo 0.5 ml in 1 injection
  Arms: Group 2

SUMMARY:
Monocentric, prospective, randomised, double-blind study of two parallel groups of 66 patients with post-reconstruction ACL hamstring contracture treated with an ultrasound-guided injection at two points on the body of the hamstring

* Group 1: botulinum toxin: 100 units (0.5ml) in 1 injection
* Group 2: placebo: 0.5 ml in 1 injection

DETAILED DESCRIPTION:
The study includes three assessments: one month after ligamentoplasty (inclusion visit) and then at M2 and M5. The therapeutic benefit of the study treatments is based on the evolution of the extension defect at M2.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient who has read and signed the consent form for participation in the study
* Patient operated on for primary ACL ligamentoplasty with or without meniscal repair
* Patient with reducible flatus >10° at 1 month post ligamentoplasty

Exclusion Criteria:

* Revision ligamentoplasty
* Multi-ligament knee
* Patient under court protection, guardianship or trusteeship
* Patient not affiliated to the French social security system
* Patient participating in another therapeutic protocol
* Pregnant woman or woman of childbearing age without effective contraception
* Patient unable to understand the informed information and/or to give written informed consent: dementia, psychosis, disturbed consciousness, non-French speaking patient
* Patient with known hypersensitivity to botulinum toxin
* Patient with peripheral neuromuscular dysfunction or pronounced atrophy of the semitendinosus muscle
* Patient treated with anticoagulants, chloroquine (or hydroxychloroquine)
* Patient treated in the previous seven days with antibiotics or muscle relaxants (such as tubocurarine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of therapeutic success, defined by the absence of extension defect at M3 post ligamentoplasty, will be compared between the groups by a Chi-2 test. | Month 2
  Therapeutic success is defined by the absence of extension defect (0 degree of flessum) at 2 months post botulinum toxin injection

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Hardy, MD, Principal Investigator — Clinique du sport
Locations (1):
- Clinique du Sport, Paris, France

IPD SHARING:
Plan to Share IPD: No